CLINICAL TRIAL: NCT06030700
Title: Multiscale RECIPES (Resilient, Equitable, and Circular Innovations With Partnership and Education Synergies) for Sustainable Food Systems (FoodImage 3; FI3) Laboratory
Brief Title: FoodImage 3 Laboratory
Acronym: FI3Lab
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Martin, Corby, K., M.D. (Individual)
Responsible Party: Principal Investigator, John Apolzan, Associate Professor-Research, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-045 B
Record Dates: First submitted 2023-08-30; First posted 2023-09-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Waste Management; Food Supply

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laboratory: Simulated kitchen setting including purchase, prep, eating and cleanout
  Interventions: Other: Controlled Conditions

INTERVENTIONS:
Other: Controlled Conditions — Use of FoodImage app to take pictures of food and/or receipts.

SUMMARY:
The Laboratory Study will be conducted at PBRC and will include participants (N=25) from a wide array of social and economic groups will be recruited and trained on the use of the FoodImage app. Participants use the app to measure food waste (including foods with inedible parts) created during a simulated meal preparation setting, a simulated meal consumption setting with plate waste, and a simulated cabinet and refrigerator clean-out of spoiled and out-of-date foods, where the number of items and the amounts of waste for each task is randomly assigned across participants and blinded from the research staff evaluating images and coding data. These participants will denote the normal discard destination (I.e., garbage, sink/disposal, feed to animal, compost) for each item as if the waste had occurred in their own home.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-65 years
* Willing to be recontacted

Exclusion Criteria:

* Refusal or unable to use an iPhone for study related purposes.
* Not willing to adhere to study procedures and study visit timelines.
* PBRC employee
* Any condition or circumstance that in the judgement of the PI could interfere with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Weight of Food Waste | At Baseline Laboratory Study Visit
  Weight (g)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data may be requested. The PI will be notified. The proposed research question must be included. All IPD that underlie results in a publication after a DTA with the institution may be provided.